CLINICAL TRIAL: NCT06888648
Title: Clinical Study to Evaluate the Safety and Efficacy of Personalized Tumor Neoantigen MRNA Therapy in Combination with PD-1 Antibody and Chemotherapy for Advanced Pancreatic Cancer.
Brief Title: Personalized Tumor Neoantigen MRNA Therapy for Advanced Pancreatic Cancer.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISPD-10
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer Metastatic; Pancreatic Cancer Non-resectable
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A (Experimental): On D1 patients start the mFOLFIRINOX every 2 weeks, and the actual number of cycles of mFOLFIRINOX will be determined by the investigators according on the patients' physical condition, disease progression, adverse effects; on the same day, started Sintilimab, 200mg, intravenous infusion, every 3 weeks; On D43 ± 3, the first efficacy assessment will be conducted. Patient with no disease progression, will continue the above treatment (mFOLFIRINOX Q2W + Sintilimab Q3W + individualized neoantigen mRNA injection Q3W); if disease progression, the patient will receive the second-line chemotherapy regimen (decided by investigators)+ Sintilimab Q3W + individualized neoantigen mRNA injection Q3W. Patients will receive efficacy assessment every 6 weeks.
  Interventions: Biological: individualized anti-tumor new antigen iNeo-Vac-R01 injection; Drug: mFOLFIRINOX Treatment Regimen; Drug: Sintilimab injection

INTERVENTIONS:
Biological: individualized anti-tumor new antigen iNeo-Vac-R01 injection — The individualized anti-tumor new antigen iNeo-Vac-R01 injection was commissioned by Hangzhou Nuanjin Biotechnology Co., Ltd., and all patients were admitted into the therapeutic intervention group. According to the results of previous non-clinical studies, the individualized mRNA injection of 100 μ g was a tolerable dose.
Drug: mFOLFIRINOX Treatment Regimen — continuous intravenous infusion of fluorouracil 2400mg / m², for 46 hours, leucovorin 400mg / m², irinotecan 135mg / m², and oxaliplatin 68mg / m², every 2 weeks
Drug: Sintilimab injection — Sintilimab Injection, 200mg, intravenous infusion, every 3 weeks

SUMMARY:
This study is a single-arm phase I/II clinical study to evaluate the effectiveness of evaluate the feasibility and safety of personalized tumor neoantigen mRNA therapy (iNeo-Vac-R01) in combination with PD-1 antibody and standard chemotherapy regimens for the treatment of patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

(1) Subjects who meet all the following entry criteria enter the pre-screening phase of the study:

1. Voluntary signing of the informed consent form;
2. Age: 18 and 75 years old, male or female;
3. Evaluation as metastatic pancreatic cancer or postoperative recurrence according to the 2024 NCCN guidelines;
4. No systemic treatment, or disease progression with gemcitabine-based first-line chemotherapy.
5. An Eastern Cooperative Oncology Group (ECOG) physical fitness status score of 0 or 1;
6. According to the efficacy evaluation criteria for solid tumors (RECIST 1.1);
7. Can obtain sufficient fresh tumor tissue samples for exome and transcriptome sequencing analysis;
8. Main organ function of heart, liver and kidney is normal:
9. Ferproductive men and women of childbearing age agree to take effective contraception from the date to the last dose of test drug; women of childbearing age included premenopause and women within 2 years after menopause;
10. Ability to follow the study protocol and follow-up procedures.

(2) Subjects who meet all the following enrollment criteria enter the formal screening stage of the study and enter the study medication process:

1. Voluntary signing of the informed consent form;
2. Age: 18 and 75 years old, male or female;
3. Pancreatic ductal adenocarcinoma (PDAC) diagnosed by pathology (histology or cytology);
4. No systemic treatment or gemcitabine-based first-line chemotherapy.
5. An Eastern Cooperative Oncology Group (ECOG) physical fitness status score of 0 or 1;
6. Main organ function of heart, liver and kidney is normal:
7. Ferproductive men and women of childbearing age agree to take effective contraception from the date to the last dose of test drug; women of childbearing age include premenopause and women within 2 years after menopause;
8. Ability to follow the study protocol and follow-up procedures.

Exclusion Criteria:

Subjects will be excluded from this study if they meet any of the following criteria:

1. Pancreatic cancer has central nervous system metastasis or meningeal metastasis;
2. At the same time with other malignant tumors, but cured basal cell cancer, thyroid cancer, cervical dysplasia, etc., have been in the disease for more than 5 years or do not considered to be easy to relapse except;
3. History of bone marrow transplantation, allogeneic organ transplantation, or allogeneic hematopoietic stem cell transplantation;
4. Patients with immunosuppressants, that is, those who require regular use of immunosuppressants 4 weeks before the screening period and the clinical study, including but not limited to the following conditions: severe asthma, autoimmune diseases or immune deficiency, treated with immunosuppressive drugs, and known history of primary immunodeficiency; except type 1 diabetes, autoimmune-related hypothyroidism requiring hormone therapy, vitiligo and psoriasis that do not require systemic therapy;
5. Active bacterial or fungal infection identified by clinical diagnosis; a history of active TB or tuberculosis;
6. Patients with positive human immunodeficiency virus (HIV) antibody, positive treponema pallidum for syphilis (TP) antibody, active hepatitis C (positive hepatitis C virus (HCV) antibody and positive HCV RNA result), active hepatitis B;
7. Herpesvirus infection (except those who scab for more than 4 weeks); respiratory virus infection (except those who have recovered for more than 4 weeks);
8. Uncontrolled complications include but are not limited to active infection, symptomatic congestive heart failure, unstable angina, arrhythmia; severe coronary artery disease or cerebrovascular disease, or other diseases considered unacceptable by the investigator;
9. Previous history of drug abuse, clinical or psychological or social factors affecting informed consent or study implementation; a history of mental illness;
10. Patients with a history of food, drug or vaccine allergy or other potential immunotherapy allergies as considered by the Investigator.
11. Women born during pregnancy or lactation;
12. The investigator is not fit for enrollment or may not complete the trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurence and frequence of AE and SAE | Up to 2 years
  Occurence and frequence of Adverse Event (AE) and Serious Adverse Event (SAE) (NCI CTCAE 5.0)

SECONDARY OUTCOMES:
Objective reponse rate (ORR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR according to RECIST1.1 criteria during the whole study
Disease control rate (DCR) | Up to 2 years
  The proportion of patients who had tumor evaluated as PR or SD according to RECIST1.1 criteria during the whole study.
Progression-free survival （PFS） | Up to 2 years
  The time from enrolled to disease pregression or death from any cause during the whole study.
Overall survival (OS) | Up to 2 years
  The time from enrolled to death from any cause during the whole study
Progression-free survival Rate（1-Y-PFS%, 2-Y-PFS%,3-Y-PFS%） | Up to 3 years
  The proportion of patients free from disease progression or death (whichever occurs first) at 12, 24, and 36 months.
Overall Survival Rate (1-Y-OS%,2-Y-OS%,3-Y-OS%) | Up to 3 years
  The percentage of patients surviving at 12, 24, and 36 months.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University Schlool of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No